CLINICAL TRIAL: NCT04458844
Title: Integrated Strength and Fundamental Movement Skill (FMS) Training in Children: a Pilot Study
Brief Title: Strength and Fundamental Movement Skill (FMS) Training in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Matthew Wright, Lecturer in Biomechanics and Strength and Conditioning, Teesside University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SSSBLRECSTUD1449
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Fundamental Movement Skill Competence
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Cluster randomised control trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fundamental Movement Skill (FMS) Training (Experimental): Exercise 2 x per week focusing on Fundamental Movement Skill Development
  Interventions: Other: Exercise
- FMS and strength (Experimental): Replacement of 50% FMS training with integrated strength training.
  Interventions: Other: Exercise
- Control (No Intervention): No intervention.

INTERVENTIONS:
Other: Exercise — Intervention programmes were designed based on previous research (Duncan, et al., 2017; Faigenbaum, et al., 2011; Miller, et al., 2006) to ensure all exercises were developmentally appropriate for the age of the participants (an example session plan can be seen in the supplementary material). Each session consisted of five activities and lasted 50 - 60 minutes. Three out of the five activities were identical for the FMS and FMS+ groups, while two differed focusing on skill development for the FMS group and strength development for the FMS+ group. The FMS and FMS+ group received their sessions twice a week for 4 weeks. The sessions were delivered at least 48 hours apart to allow recovery and to reduce the risk of fatigue effecting performance (Faigenbaum, et al., 1996). All sessions were led by a researcher and a qualified sports coach.
  Arms: FMS and strength; Fundamental Movement Skill (FMS) Training

SUMMARY:
Competence in Fundamental movement skills (FMS) is essential to enable children to be physical active. The aim of this study was to investigate the effects of integrated FMS skill training (balancing and stabilisation skills, locomotor skills [e.g. run, hop, jump, crawl] and object control / manipulation [e.g. dribbling, rolling, striking, kicking and catching i.e. a ball] with strength training on FMS performance in children.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 - 11 years in a participating primary school (cluster) for which the Head Teacher has provided consent.
* Parental consent received

Exclusion Criteria:

* No parental consent

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-07-22 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Change in product-process assessment of FMS via the Canadian agility and movement skills assessment (CAMSA) | Baseline data was collected mid-June 2018 at the primary schools, one week prior to the intervention. Post testing data collection was in the week immediately after the final week of the four week intervention.
  The Canadian agility and movement skills assessment (CAMSA), which combines product- and process-oriented outcomes was used to assess FMS. Full details of the CAMSA can be found in the Canadian Assessment of Physical Literacy Manual, 2017. Briefly, the CAMSA requires participants to travel a total distance of 20m while completing seven different movement skill tasks (Longmuir et al 2017) around an agility style course. Process oriented criteria were used to assess the performance of each movement skill. In addition, the throw and kick were scored as either hitting or missing a target 5m away (product assessment). Finally, the overall time taken to complete the course was recorded (product assessment) and converted into a timed score using pre-defined time criteria scores. The CAMSA raw score was calculated by adding the individual skill scores (max of 14 points) and the time criteria score (max of 14 points) giving an individual score between 1 and 28 points.

SECONDARY OUTCOMES:
Change in product assessment of FMS | Baseline data was collected mid-June 2018 at the primary schools, one week prior to the intervention. Post testing data collection was in the week immediately after the final week of the four week intervention.
  The investigators assessed locomotor performance through a countermovement jump and sprint assessments. Jump height was calculating from flight time measured by the Optojump Next (Microgate, Italy). Children were allowed up to three trial repetitions before completing three maximal jumps with the best performance used for analysis. Jumps were not counted if the children tucked their legs in the air or landing outside of the 1m square testing area. Sprint times were recorded over a distance of 40m to the nearest 0.01 second using an infrared timing gate system (Brower timing systems, Draper, USA). Sprints were repeated three times and the best score taken for analysis.
Change in strength | Baseline data was collected mid-June 2018 at the primary schools, one week prior to the intervention. Post testing data collection was in the week immediately after the final week of the four week intervention.
  Grip strength (Takei Grip-D) and counter movement jump (CMJ) (Optojump Next, Microgate, Italy) were recorded as measures of upper and lower body strength, respectively. The children followed a set of standardised instructions and completed three attempts on each test to give an average score for each test.

CONTACTS AND LOCATIONS:
Locations (1):
- Teesside University, Middlesbrough, England, United Kingdom